CLINICAL TRIAL: NCT00744796
Title: Early Experience With Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK) in Patients With Corneal Endothelial Cell Dysfunction: Clinical Outcomes and Diagnostic Imaging Analysis
Brief Title: Early Experience With Descemet's Stripping Automated Endothelial Keratoplasty
Acronym: DSAEK
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, V. Vinod Mootha, Faculty Sponsor, University of Texas Southwestern Medical Center
Other Study IDs: 102006-017
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Corneal Edema Secondary to Corneal Endothelial Dystrophy
Keywords: Endothelial Dystrophy; Fuchs' Endothelial Corneal Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DSAEK: Outcomes in patients with corneal edema: Best spectacle corrected visual acuity and anterior segment optical coherence tomography (OCT) at minimum will be performed in patients who have undergone DSAEK for corneal edema secondary to corneal endothelial dysfunction.
  Interventions: Procedure: DSAEK; Diagnostic Test: Anterior Segment Optical Coherence Topography (OCT); Diagnostic Test: Best Spectacle Corrected Visual Acuity (BSCVA)

INTERVENTIONS:
Procedure: DSAEK — Endothelial Keratoplasty
Diagnostic Test: Anterior Segment Optical Coherence Topography (OCT) — Non-contact, high resolution, cross sectional imaging of the anterior segment of the eye.
Diagnostic Test: Best Spectacle Corrected Visual Acuity (BSCVA) — Visual acuity determined using a combination of detecting hand motion, counting fingers displayed and reading Snellen charts at specific distances.

SUMMARY:
The purpose of this study is to report the early clinical outcomes in patients undergoing Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK) for corneal edema secondary to corneal endothelial cell dysfunction, and to correlate this clinical data with the latest generation of imaging modalities available for the anterior segment.

DETAILED DESCRIPTION:
A concurrent study for retrospective as well as prospective cases of patients undergoing DSAEK procedures for indication of corneal endothelial cell dysfunction. For the retrospective study, all cases of DSAEK procedures performed at UT-Southwestern for corneal edema secondary to endothelial cell dysfunction will be considered. The clinical outcomes of these surgeries will be analyzed and correlated with the anterior segment imaging from each case. Statistical analysis will then be performed on the data collected. For the prospective arm of this trial, we propose to recruit up to 200 current patient cases of corneal edema second corneal endothelial cell dysfunction. These patients will undergo ocular imaging studies in addition to routine ocular exams performed before surgery and at the discretion of the investigational physician at 3 to 6-months and 6 to 9-months after surgical treatment. Various imaging modalities would include corneal topography, pentacam, anterior segment OCT, wavefront measurement and Tandem Scanning Confocal Microscopy (TSCM). The patients who have already had the DSAEK procedure done in the past will undergo ocular examination as well as various imaging studies at their post op follow up visits. All these modalities are routinely used as standard of care practice and are non-invasive. The data from the ocular examination and various imaging techniques will be pooled and analyzed at the end of the study in order to identify the factors that influence the visual outcome. We believe this will help us learn more about this interesting and innovative technique while at the same time help us improve the method further in order to obtain better results in future patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and up, where any age over 89 will be recorded as 'greater than 89', who have reviewed and understood the study consent form will be invited to participate in this study.
* They will be recruited based on diagnosis of corneal edema secondary to endothelial cell dysfunction undergoing DSAEK either alone or in conjunction with phacoemulsification and intraocular lens implantation at the University of Texas Southwestern Medical Center at Dallas.

Exclusion Criteria:

* Patients younger than 18 years will not be considered for this trial.
* The study will include all patients (no exclusion criteria) who have undergone and will undergo DSAEK implantation for corneal edema secondary to corneal endothelial dystrophy with an effort to determine its success.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients 18 years or older with a clinical diagnosis of corneal edema secondary to endothelial cell dysfunction undergoing DSAEK either alone or in conjunction with phacoemulsification and intraocular lens implantation at the University of Texas Southwestern Medical Center between May, 2006 and July, 2007.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Mootha, MD, Principal Investigator — UTSW Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center - Aston Ambulatory Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty one patients from UT Southwestern Medical Center's Ophthalmology clinic were included.
Groups:
- DSAEK Group: Patients who have corneal dystrophy and have elected to have DSAEK performed on his/her eye(s).
Period: Pre-operative
Arm/Group | DSAEK Group
Started | 21
Completed | 21
Not Completed | 0
Period: Post-Operative Day 1
Arm/Group | DSAEK Group
Started | 21
Completed | 21
Not Completed | 0
Period: Post-Operative 3-6 Months
Arm/Group | DSAEK Group
Started | 21
Completed | 21
Not Completed | 0
Period: Post-Operative 6-9 Months
Arm/Group | DSAEK Group
Started | 21
Completed | 9
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | DSAEK Group
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants] — Participants in Study
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 17
Sex/Gender, Customized [Count of Participants; unit: Participants] — Collecting the gender information amongst all participants.
  Participants
    Female | 9
    Male | 12
Best-Spectacle Corrected Visual Acuity (BSCVA) [Count of Participants; unit: Participants] — Detection of hand motion, counting of fingers displayed and Snellen chart reading accuracy were used.
  Participants
    Snellen fraction < or = 20/200 | 0
    Snellen fraction < or = 20/50 and >20/200 | 5
    Snellen fraction < or = 20/20 and >20/50 | 12
    Hand Motion only | 1
    Finger Count only | 3

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle Corrected Visual Acuity (BSCVA)
Description: Best spectacle corrected visual acuity determined using detection of hand motion, counting of displayed fingers and accuracy of Snellen chart reading at specified distances.
Time Frame: 6-9 months Post-Operative
Population: The number of participant, for analysis, were determined per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | DSAEK Group
Number analyzed (Participants) | 21
Participants
  hand motion only | 1
  finger count only | 3
  Snellen fraction < or = 20/200 | 7
  Snellen fraction < or = 20/50 and >20/200 | 9
  Snellen fraction < or = 20/20 and >20/50 | 1

2. Primary Outcome: Central Corneal Thickness
Description: The central corneal thickness was determined manually by a single investigator from optical coherence tomography (OCT) measurements. A horizontal cross-sectional image with good central reflective light representing the anterior corneal vertex was used.
Time Frame: 6 to 9 Months Post-Operative
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | DSAEK Group
Number analyzed (Participants) | 21
micrometer | 686.6 (72)

3. Primary Outcome: Peripheral Corneal Thickness
Description: Peripheral corneal thickness was determined manually by a single investigator using the mean of 2 measurements taken by OCT 3.5 mm from the center of the cornea.
Time Frame: 6 to 9 Months Post-Operative
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | DSAEK Group
Number analyzed (Participants) | 21
micrometer | 710 (105)

ADVERSE EVENTS:
Arm/Group | DSAEK Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes